CLINICAL TRIAL: NCT06389266
Title: Network-Targeted Neuromodulation for Nicotine Dependence in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Heather Burrell Ward, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 221550
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Nicotine Dependence
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All participants receive five days of DMN-targeted cTBS and five days of L DLPFC-targeted iTBS. The order in which participants receive the two types of TMS is randomized.
Masking Description: The study is not sham-controlled, as both arms are active TMS treatments. The type of TMS is not masked from the participant or the investigator. Statistician will be blinded to intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- L DLPFC-Targeted iTBS, Then DMN-Targeted cTBS (Active Comparator): Participants will first receive intermittent theta burst stimulation (iTBS) at 100% active motor threshold (AMT) anatomically targeted to the left dorsolateral prefrontal cortex for five consecutive days. iTBS will be administered in a pattern consisting of 2s trains of 3 pulses at 50Hz, repeated at 5Hz, every 10s for a total of 600 pulses. There will then be a washout period of at least two weeks before starting the DMN-Targeted cTBS. Participants will then receive continuous theta burst stimulation (cTBS) at 100% AMT targeted to an individual-specific map of the left parietal node of the default mode network for five consecutive days. cTBS will be administered in a pattern consisting of 1 60s train of 3 pulses at 50Hz, repeated at 5Hz, for a total of 600 pulses.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- DMN-Targeted cTBS, Then L DLPFC-Targeted iTBS (Active Comparator): Participants will first receive continuous theta burst stimulation (cTBS) at 100% AMT targeted to an individual-specific map of the left parietal node of the default mode network for five consecutive days. cTBS will be administered in a pattern consisting of 1 60s train of 3 pulses at 50Hz, repeated at 5Hz, for a total of 600 pulses. There will then be a washout period of at least two weeks before starting the L DLPFC-Targeted iTBS. Participants will receive intermittent theta burst stimulation (iTBS) at 100% active motor threshold (AMT) anatomically targeted to the left dorsolateral prefrontal cortex for five consecutive days. iTBS will be administered in a pattern consisting of 2s trains of 3 pulses at 50Hz, repeated at 5Hz, every 10s for a total of 600 pulses.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows the selective external manipulation of neural activity in a non-invasive manner. During TMS, a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field that in turn induces electrical current in neurons and allows the modulation of neural circuitry. The combination of rTMS with functional magnetic resonance imaging allows the selective targeting and modulation of brain networks. The repeated application of rTMS can cause long term changes in behavior and task performance that is reflected in altered brain network connectivity.

SUMMARY:
The goal of this clinical trial is to compare two active types of transcranial magnetic stimulation in two nicotine-using populations: nicotine-using people with psychosis and nicotine-using people without a diagnosis of a psychotic disorder. The main questions it aims to answer are:

1. Can rTMS change functional connectivity in brain circuits associated with nicotine use?
2. Are those rTMS-induced changes in functional connectivity related to craving?

Participants will complete tasks assessing their cognitive performance and craving before and after each week of TMS. Researchers will compare the effect of each TMS intervention on participants with and without psychosis to see if one type of TMS has an effect on nicotine craving.

DETAILED DESCRIPTION:
This study proposes to test the hypothesis that the brain circuits most relevant to nicotine use in schizophrenia are distinct from pathways identified in nicotine-using people without psychosis. This study seeks to provide evidence that targeted stimulation of the Default Mode Network (DMN) leads to both altered network activity and a concomitant behavioral change in cue-induced craving and cognitive performance in individuals with schizophrenia and schizoaffective disorder, while targeted stimulation of the left dorsolateral prefrontal cortex (L DLPFC) leads to these changes in nicotine-using people without psychosis.

The investigators will test this hypothesis in a crossover design comparing 1) DMN-targeted continuous theta burst stimulation (cTBS) and 2) L DLPFC-targeted intermittent theta burst stimulation (iTBS). cTBS and iTBS are types of rTMS. cTBS has inhibitory effects and reduces functional connectivity, while iTBS is excitatory and increases connectivity (Huang et al. 2005). By applying cTBS to the DMN, a target that modulates craving in schizophrenia, the investigators expect DMN connectivity to decrease, thereby decreasing craving. Excitatory stimulation (e.g. iTBS) to the L DLPFC reduces craving in smokers without psychosis (Tseng et al. 2022).

This study will test a model that integrates brain network pathophysiology and cognition to 1) explain the prevalence of nicotine use in schizophrenia and 2) identify a target for engagement in schizophrenia. This study seeks to establish a neuroscientific framework to guide future treatment-oriented studies aimed at reducing craving and improving cognitive performance in individuals with schizophrenia and schizoaffective disorder.

Aim 1: Target Engagement: Determine if rTMS manipulates functional connectivity of each target (DMN, L DLPFC) (n=60). Hypothesis 1A: Functional connectivity of the entire DMN will decrease after 5 days of DMN-targeted cTBS. Hypothesis 1B: Functional connectivity of the L DLPFC to the left insula will increase after 5 days of L DLPFC-targeted iTBS. As an exploratory hypothesis, the investigators will test if there is an effect of diagnosis on connectivity change.

Aim 2: Clinical Efficacy: Determine if rTMS affects cue-induced craving and if craving change correlates with change in functional connectivity (n=60). Hypothesis 2A: Both DMN-targeted and L DLPFC-targeted rTMS will significantly reduce craving. Hypothesis 2B: Craving change will be correlated with functional connectivity change. As an exploratory hypothesis, in individuals with schizophrenia, DMN-targeted cTBS will be more efficacious than L DLPFC-targeted iTBS.

Aim 3: Determine if individual differences in rTMS-induced network connectivity change are explained by individual differences in network controllability (n=60). There is significant heterogeneity in individual response to rTMS, even with network-targeted approaches. This may be related to network controllability, a metric of the average input energy required to change brain state (Bassett and Sporns 2017). It is critical to understand predictors of network change for optimal rTMS target selection in clinical trials. Hypothesis 3: Individual differences in rTMS-induced change in DMN connectivity will be associated with average controllability of the DMN rTMS stimulation site.

ELIGIBILITY:
Inclusion Criteria for Participants with Psychosis:

* Age between 18-65 years
* Diagnosis of either schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual for Mental Disorders (DSM-5) criteria and confirmed by Structured Clinical Interview for the DSM (SCID) (First et al. 2015)
* Current nicotine use (confirmed by expired carbon monoxide or urine cotinine)
* Must be able to read, speak and understand English
* Must be judged by study staff to be capable of completing the study procedures
* Participants will be in stable outpatient psychiatric treatment and psychiatrically stable with no recent (within the past 90 days) psychiatric hospitalizations or changes in their psychiatric medication regimens.

Inclusion Criteria for People without Psychosis:

- All of the above except for participants will not have a diagnosis of schizophrenia or schizoaffective disorder nor a first-degree relative with a psychotic disorder.

Exclusion Criteria for All Participants:

* DSM-5 intellectual disability
* Substance use disorder (other than nicotine) within the past three months Positive urine drug screen for illicit substance use that can increase seizure risk (cocaine, benzodiazepines, amphetamine, methamphetamine)
* Any history of a progressive or genetic neurologic disorder (e.g. Parkinson's disease, multiple sclerosis, tuberous sclerosis, Alzheimer's Disease) or acquired neurological disease (e.g. stroke, traumatic brain injury, tumor), including intracranial lesions
* History of head trauma resulting in any loss of consciousness (>15 minutes) or neurological sequelae
* Current history of poorly controlled headaches including chronic medication for migraine prevention
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* Any metal in the brain or skull (excluding dental fillings) or elsewhere in the body unless cleared by the responsible covering MD (e.g. MRI compatible joint replacement)
* Any devices such as pacemaker, medication pump, nerve stimulator, transcutaneous electrical nerve stimulation (TENS) unit, ventriculo-peritoneal shunt unless cleared by the responsible covering MD
* All female participants of child-bearing age will be required to have a pregnancy test; any participant who is pregnant or planning to become pregnant will not be enrolled in the study
* Medications will be reviewed by the responsible covering physician and a decision about inclusion will be made based on the participant's past medical history, drug dose, history of recent medication changes or duration of treatment, and use of central nervous system (CNS) active drugs. The published TMS guidelines review of medications to be considered with rTMS will be taken into consideration given their described effects on cortical excitability measures.
* Any changes in medications or hospitalizations within the past 90 days.
* Participants who, in the investigator's opinion, might not be suitable for the study or would be unable to tolerate the study visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Resting-state functional connectivity | Baseline to one week, and three weeks to five weeks
  The investigators will evaluate the effect of DMN-targeted cTBS on functional connectivity of the left parietal node of the DMN and the entire default mode network. The investigators will also evaluate the effect of L DLPFC-targeted iTBS on functional connectivity of the L DLPFC.
Cue-induced craving | Baseline to one week, and three weeks to five weeks
  The investigators will evaluate the effect of DMN-targeted cTBS and L DLPFC-targeted iTBS on self-reported craving before and after presentation of visual nicotine cues. Craving is measured on a scale from 0 to 10, with 10 being the highest level of craving.
Tiffany Brief Questionnaire of Smoking Urges (QSU) | Baseline to one week, and three weeks to five weeks
  The investigators will evaluate the effect of DMN-targeted cTBS and L DLPFC-targeted iTBS on QSU scores. The QSU-Brief has a range of 10-70, with higher scores indicating higher smoking urges.
Self-reported craving | Baseline to one week, and three weeks to five weeks
  The investigators will evaluate the effect of DMN-targeted cTBS and L DLPFC-targeted iTBS on self-reported craving, measured by a Visual Analog Scale of nicotine craving. Craving is measured on a scale from 0 to 10, with 10 being the highest level of craving.

SECONDARY OUTCOMES:
Wisconsin Smoking Withdrawal Scale (WSWS) | Baseline to one week, and three weeks to five weeks
  The investigators will evaluate the effect of DMN-targeted cTBS and L DLPFC-targeted iTBS on self-reported withdrawal symptoms.The WSWS has a range of 0-112, with higher scores indicating higher withdrawal.
Fagerstrom Test for Nicotine Dependence (FTND) | Baseline to one week, and three weeks to five weeks
  The investigators will evaluate the effect of DMN-targeted cTBS and L DLPFC-targeted iTBS on nicotine dependence severity. The FTND has a range of 0-10, with higher scores indicating greater nicotine dependence.
Self-reported nicotine use | Baseline to one week, and three weeks to five weeks
  The investigators will evaluate the effect of DMN-targeted cTBS and L DLPFC-targeted iTBS on self-reported nicotine use, measured by the Timeline Follow Back and the Recent Substance Use Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Heather B Ward, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Tseng PT, Zeng BS, Hung CM, Liang CS, Stubbs B, Carvalho AF, Brunoni AR, Su KP, Tu YK, Wu YC, Chen TY, Li DJ, Lin PY, Hsu CW, Chen YW, Suen MW, Satogami K, Takahashi S, Wu CK, Yang WC, Shiue YL, Huang TL, Li CT. Assessment of Noninvasive Brain Stimulation Interventions for Negative Symptoms of Schizophrenia: A Systematic Review and Network Meta-analysis. JAMA Psychiatry. 2022 Aug 1;79(8):770-779. doi: 10.1001/jamapsychiatry.2022.1513. PMID 35731533
- [Background] Bassett DS, Sporns O. Network neuroscience. Nat Neurosci. 2017 Feb 23;20(3):353-364. doi: 10.1038/nn.4502. PMID 28230844

DOCUMENTS (1):
  • Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT06389266/ICF_000.pdf